CLINICAL TRIAL: NCT04898764
Title: Characterisation and Intervention Study in Patients With Long-term Use of Nasal Decongestants
Brief Title: Research on Underlying Causes of Long-term Use of Nasal Decongestants and the Structured Withdrawal of the Decongestant
Acronym: Momestasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO/2019/005; 2019-003254-91 (EudraCT Number)
Record Dates: First submitted 2020-10-16; First posted 2021-05-24 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Rhinitis Medicamentosa
Keywords: non-allergic drug-induced rhinitis
MeSH Terms: interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (No Intervention): This study arm will only participate in part A of the study (Characterisation study) and thus will not receive the study drug. A maximum of 35 healthy volunteers will be included in this study arm.
- Patients with long-term use of nasal decongestants (Experimental): A maximum of 100 patients with long-term use of nasal decongestants will be included in this study arm, for part A of the study (Characterisation study).
  The investigators will consecutively recruit patients from part A (Characterisation study) into part B of the study (Intervention study) until a total of 35 patients completed all study-related visits of part B. During the intervention study, patients with long-term use of nasal decongestants will administer Mometasone furoate intranasally, two doses (50µg/actuation) in each nostril, twice daily (total daily dose of 400µg) during a 12 week period.
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Mometasone Furoate — Mometasone furoate nasal spray suspension, 50µg/actuation
  Arms: Patients with long-term use of nasal decongestants

SUMMARY:
Rhinitis medicamentosa (RM) is a form of non-allergic medication-induced rhinitis characterised by nasal congestion. This nasal congestion is the result of the overuse of intranasal decongestants which leads to rebound congestion when the medication wears off. This prompts the user of the nasal decongestant to administer more in order to obtain relief from the feeling of a blocked nose. Therefore, the patient ends up in a vicious cycle caused and temporarily relieved by the use of medication.The diagnosis of rhinitis medicamentosa depends greatly on the history of prolonged use of the nasal decongestant, since real diagnostic criteria have not yet been established. It is unclear if these patients suffer from an underlying (undetected and/or untreated) nasal condition which might have caused the patient to start using the nasal decongestant in the first place. Therefore, the aim of the first part of this study (Part A) is to characterize patients with long-term use of nasal decongestants to examine if an underlying nasal condition is present. The investigators will include healthy volunteers in part A of the study to be able to compare their test results with those of patients with long-term use of nasal decongestants and hence be able to detect differences.

Thus far, the treatment of RM has been the topic of debate. Several treatment regimens have been proposed in literature, but most study authors agree that it is essential to stop the overuse of the nasal decongestant either immediately or gradually to limit withdrawal symptoms. For this part of the study (Part B: intervention study), the investigators aim to reduce the long-term use of nasal decongestants based on a structured withdrawal programme comprising medication (nasal corticosteroid spray) and motivational interviewing. Only patients with long-term use of nasal decongestants are eligible to participate in this part of the study. They will be rescreened prior to inclusion into this part of the study.

DETAILED DESCRIPTION:
The study comprises two parts:

* Part A: Characterisation study (both healthy volunteers and patients with long-term use of nasal decongestants)
* Part B: Intervention study (only patients with long-term use of nasal decongestants). Patients will be rescreened prior to inclusion into part B of the study. Participants will receive the intervention (Mometasone furoate nasal spray) during a 12-week period

Part A (characterisation study) consists of three study-related contact moments:

1. Screening visit
2. Telephone contact
3. Ear-, nose- and throat examination (actual characterisation study)

Part B (intervention study) consists of five contact moments:

1. Start-up of the intervention
2. Telephone contact (during follow-up 1 period)
3. Follow-up 1 (After 6 weeks of intervention*)
4. Follow-up 2 (After 12 weeks of intervention*)
5. Telephone follow-up (6 months post start-up of the intervention*) * Study windows foreseen in the protocol

Procedures performed during part A of the study:

* Peak Nasal Inspiratory Flow (PNIF) measurements
* Nasal endoscopy
* Collection of blood samples and nasal secretions
* Completion of questionnaires
* Completion of patient diary
* Collection of data regarding medication use
* Skin prick testing
* Completion of patient diary
* Medical photography of the face and nose
* Telephone follow-up

Procedures performed during part B of the study:

* Urine pregnancy test
* Collection of data regarding medication use
* Counselling conversations with the researchers
* Completion of questionnaires
* Completion of patient diary
* Drug accountability
* Daily administration of Mometasone furoate (by the patients themselves, during a 12 week period)
* PNIF measurements
* Nasal endoscopy
* Collection of blood samples and nasal secretions
* Telephone follow-up

ELIGIBILITY:
Inclusion Criteria Healthy Volunteers (only included in part A of the study):

* Aged 18 years or older
* Sufficient knowledge of the Dutch language

Exclusion Criteria Healthy Volunteers (only included in part A of the study):

* Subjective presence of nasal disease (i.e. the study subject indicates to experience any nasal symptoms, an occasional common cold not taken into account)
* Established diagnosis of a nasal disorder (e.g. allergy, nasal polyps, …) or a positive allergy test (skin prick test or blood test)
* Prior nasal surgery
* Asthma
* Use of an oral corticosteroid in the month prior to the screening visit
* Significant disease(s) that might interfere with the study, based on the judgement of the investigator
* Current use of a nasal decongestant, more than two episodes of 7 days use of a nasal decongestant in the previous year or less than two episodes of 7 days use (in the previous year) but last use less than a month prior to the screening visit
* Other medication used to treat nasal symptoms (intranasal corticosteroids, oral or intranasal antihistamines, oral decongestants …)
* History of rhinitis medicamentosa (either patient-reported long-term use of a nasal decongestant or a diagnosis of rhinitis medicamentosa)
* Pregnancy, trying to become pregnant (during the duration of the study) or breastfeeding

Inclusion Criteria patients with long-term use of nasal decongestants: part A:

* Aged 18 years or older
* Daily use of a nasal decongestant for at least 6 months. Following ATC-codes are considered, when the spray or drops contain a nasal decongestant and the drug is thus intended for short-term use only: R01AA, R01AB, R01AD52, R01AD53
* Sufficient knowledge of the Dutch language

Exclusion Criteria patients with long-term use of nasal decongestants: part A:

* Pregnancy, trying to become pregnant (during the duration of the study) or breastfeeding
* Use of an oral corticosteroid in the month prior to the screening visit
* Use of an oral decongestant in the week prior to the screening visit
* Significant disease(s) that might interfere with the study, based on the judgement of the investigator

Inclusion Criteria patients with long-term use of nasal decongestants: part B:

* Aged 18 years or older
* Daily use of a nasal decongestant for at least 6 months.Following ATC-codes are considered, when the spray or drops contain a nasal decongestant and the drug is thus intended for short-term use only: R01AA, R01AB, R01AD52, R01AD53
* Sufficient knowledge of the Dutch language

Exclusion Criteria patients with long-term use of nasal decongestants: part B:

* Pregnancy, trying to become pregnant (during the duration of the study) or breastfeeding
* Glaucoma
* Use of an oral corticosteroid in the month prior to the start of the intervention
* Use of an oral decongestant in the week prior to the start of the intervention
* Significant disease(s) that might interfere with the study, based on the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of study subjects with long-term use of nasal decongestants able to completely withdraw the use of the nasal decongestant after 12 weeks of intervention. | Assessed at follow-up 2 (12 weeks post start up intervention)
  To evaluate the effectiveness of a standardized, structured withdrawal plan based on Mometasone furoate combined with motivational interviewing to reduce the overuse of nasal decongestants.
  For this study, complete withdrawal is defined as at least 7 consecutive days without any use of a nasal decongestant.
Proportion of study subjects who were able to completely withdraw the long-term use of nasal decongestants at follow-up 2 (after 12 weeks of intervention) who relapsed by the time of follow-up 3 (6 months after the start-up of the intervention). | Assessed at follow-up 3 (6 months post start-up of the intervention)
  To evaluate the relapse rates of patients with former nasal decongestant overuse. For this study, relapse is defined as daily use of a nasal decongestant for more than 7 consecutive days after prior full withdrawal of the nasal decongestant

SECONDARY OUTCOMES:
Change from intervention baseline (part B) to week 12 of intervention in Rhinitis Control Assessment Test (RCAT) score (RCAT scores range from 6 to 30, with higher scores indicating greater rhinitis symptom control) | Assessed at intervention baseline, follow-up 1 (6 weeks post start-up intervention), and follow-up 2 (12 weeks post start-up intervention)
  To evaluate the change in rhinitis control due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in home measured PNIF as captured in diary on a fixed day every week | Assessed during screening period (2 weeks) and intervention period (12 weeks post start up intervention) on a weekly basis
  To evaluate the change in nasal patency due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in hospital measured Peak Nasal Inspiratory Flow (PNIF) | Assessed at intervention baseline, follow-up 1 (6 weeks post start-up intervention), and follow-up 2 (12 weeks post start-up intervention)
  To evaluate the change in nasal patency due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in Visual Analogue Scale (VAS) for nasal obstruction. Range 0mm - 100mm with higher values indicating worse outcome | Assessed at intervention baseline, follow-up 1 (6 weeks post start-up intervention), and follow-up 2 (12 weeks post start-up intervention)
  To evaluate the change in nasal patency due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in Visual Analogue Scale (VAS) for nasal symptoms (nasal obstruction, runny nose, sneezing) as captured in the daily diary. Range 0mm-100mm with higher values indicating worse outcome | Assessed during screening period (2 weeks) and intervention period (12 weeks) on a daily basis
  To evaluate the change in nasal patency due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in Mini Rhinoconjunctivitis Quality of Life Questionnaire (miniRQLQ) (14 items, 0= no impairment to 6= severely impaired; higher scores indicate greater impairment of QoL) | Assessed at intervention baseline, follow-up 1 (6 weeks post start-up intervention), and follow-up 2 (12 weeks post start up intervention)
  To evaluate the change in disease specific health-related quality of life (HRQoL) due to the withdrawal of the nasal decongestant
Change from intervention baseline (part B) to week 12 of intervention in PROMIS Sleep Disturbance Short form 8b scores (Raw scores range from 8 to 40, with higher scores indicating greater sleep disturbance) | Assessed at intervention baseline, follow-up 1 (6 weeks post start-up intervention), and follow-up 2 (12 weeks post start-up intervention)
  To evaluate the change in sleep disturbance due to the withdrawal of the nasal decongestant
Change from baseline (part A) to week 12 of intervention in nasal endoscopy outcomes, assessed with our newly developed nasal endoscopy scoring sheet (containing Visual Analogue Scales (0-100mm), a colour scale and a nasal polyp scoring system) | Assessed at baseline (characterisation study) and at follow-up 2 (12 weeks post start-up intervention)
  To evaluate the change in nasal endoscopy outcomes due to the withdrawal of the nasal decongestant

OTHER OUTCOMES:
Change from baseline (part A) to week 12 of intervention in exploratory biomarkers of inflammation and immune response in blood samples and nasal secretions (multiplex analysis of cytokines) | Assessed at baseline (characterisation study) and at follow-up 2 (12 weeks of intervention)
  To assess the effect of withdrawal on exploratory biomarkers of inflammation and immune response in blood samples and nasal secretions

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gevaert, MD, PhD, Principal Investigator — Ghent University Hospital, Ghent, Belgium
Locations (1):
- Ghent University Hospital, Ghent, Belgium